CLINICAL TRIAL: NCT06129396
Title: Effects of Aerobic Exercise Intervention in Adolescents With Attention-deficit/Hyperactivity Disorder (ADHD)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 202211047RIND
Record Dates: First submitted 2023-10-31; First posted 2023-11-13 (Actual); Last update posted 2023-11-13 (Actual); Status verified 2023-10

CONDITIONS: Attention Deficit Hyperactivity Disorder
Keywords: Attention Deficit Hyperactivity Disorder; A single bout of aerobic exercise; Executive functions; Neurophysiology
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Aerobic exercise group (Experimental): The aerobic exercise consists of: (1) 5 min warm-up exercise, (2) 20 min aerobic exercise with heart rate (HR) at target zone (one research assistant will be onsite to monitor whether the HR is around the range of moderate intensity), and (3) 5 min cool-down exercise.
  Interventions: Other: Aerobic exercise
- Video-watching group (Active Comparator): The video-watching group will be asked to watch a nature documentary for 30 mins
  Interventions: Other: Video-watching

INTERVENTIONS:
Other: Aerobic exercise — The aerobic exercise consists of: (1) 5 min warm-up exercise, (2) 20 min aerobic exercise with HR at target zone (one research assistant will be onsite to monitor whether the HR is around the range of moderate intensity), and (3) 5 min cool-down exercise.
  Arms: Aerobic exercise group
Other: Video-watching — The video-watching group will be asked to watch a nature documentary for 30 mins
  Arms: Video-watching group

SUMMARY:
The goal of this clinical trial is to investigate the neurophysiological foundation of the impact of the acute effects of controlled aerobic exercise intensity in adolescents with ADHD, its involvement in cognitive processes, and clinical outcomes in respect to executive functions.

The main questions it aims to answer are:

* To find out the effects of a single bout of aerobic exercise intervention on neurophysiology and executive functions in adolescents with ADHD
* To examine the relationship between neurophysiology and executive functions following a single bout of aerobic exercise intervention

Participants will be asked to do three different executive function tasks regarding inhibitory control, working memory and cognitive planning and receive the evaluation of motor cortex excitability via transcranial magnetic stimulation (TMS) before and after a single bout of 30-min aerobic cycling exercise of moderate intensity. Researchers will compare the control group with 30-min video-watching to see if effects of a single bout of aerobic exercise intervention on neurophysiology and executive functions in adolescents with ADHD.

DETAILED DESCRIPTION:
Attention-deficit hyperactivity disorder (ADHD) is the most prevalent neuropsychiatric disorders affecting 5-10% of children worldwide (7~8% in Taiwan) characterized by a persistent pattern of inattention and/or hyperactivity/impulsivity. Recent survey estimated that around 57% of children with ADHD will continue to have persistent symptoms into adolescents and adulthood. Due to the dynamic neurocognitive development process, and the transition and formation of educational and social relationship, adolescents (13-17 years) represent critical periods in the phase of life. Emerging literature has proposed the main conditions of ADHD are related to cognitive function impairments such as inhibitory control, working memory and cognitive planning. These deficits disrupt educational process, harm academic and social functions, and seriously reduce quality of life for adolescents with ADHD.

Recently, noninvasive brain stimulation techniques are considered for investigating the neural mechanism of neurodevelopmental disorders including ADHD. Previous studies using transcranial magnetic stimulation (TMS) in combination with motor-evoked potentials (MEPs; muscle contraction in response to TMS) have reported deficits in specific inhibitory functions of the motor loop in ADHD. In line with this, our previous study found decreased intracortical inhibition and enhanced intracortical facilitation in ADHD subjects compared to healthy control (under review). These findings implied that ADHD causes stem from disturbances in large-scale brain networks Therefore, it is essential to understand the neurophysiological mechanism in ADHD, and furthermore develop effective interventions based on this foundation.

Aerobic exercise has been suggested as a safe and low-cost adjunctive therapy for ADHD and is known to have beneficial effects on cognition and behavioral performance in children and adolescents. The underlying mechanism depends at least partially on mechanisms of neuroplasticity. Animal data suggest that neuronal excitability is enhanced by aerobic exercise via suppressing gamma-aminobutyric acid (GABA)-ergic inhibition and facilitating the activation of N-methyl-D-aspartate (NMDA) receptors. Furthermore, aerobic exercise enhanced the induction of long-term potentiation (LTP) which is thought to play a key role in the cellular mechanisms of learning and memory. These findings align with human data. Our and other studies have shown that aerobic exercise can enhance cortical excitability via increasing intracortical facilitation and reducing inhibition in healthy subjects by TMS. At the cognitive domain, animal models have shown that aerobic exercise prominently affects diverse cognitive functions, including learning and memory. Similarly, in the human study, a single bout of light-intensity aerobic exercise promotes performance of a visuomotor accuracy-tracking task and verbal memory. Meta-analytic research has shown beneficial effects of moderate to vigorous-intensity aerobic exercise on cognitive performance in humans. Specific for ADHD population, previous results showed significant improvement in inhibitory control, speed of processing, and attention after acute aerobic exercise (30 mins cycling: a 5 min warm up, 20 min of core exercise, and a 5 min cool-down) at moderate intensity. Taken together, these studies suggest that impact of aerobic exercise might not restricted to motor domain. Additionally, the positive effects of aerobic exercise on cognitive processes and clinical outcomes might be caused by its mediating effects on neural mechanisms.

According to our research experienced, we are interested in the neurophysiological foundation of the impact of the acute effects of controlled aerobic exercise intensities in adolescents with ADHD, its involvement in cognitive processes, and clinical outcomes. Combined application of neurophysiological recording tools, including non-invasive brain stimulation, are suited to explore the impact of aerobic exercise on cortical physiology of motor and prefrontal cortex, and the functional association of cognition and clinical performance in humans. We will apply TMS to obtain evoked potentials recorded either with electromyography (EMG) or EEG to cortical excitability, also with regard to the contributions of specific transmitters and neuromodulators, such as glutamate and GABA, over task-relevant target areas such as motor and prefrontal cortex. Furthermore, we will combine cognitive task (e.g., inhibitory control, working memory and cognitive planning tasks) to explore the association between the neurophysiological effects of aerobic exercise and respective cognitive and clinical alterations. The study will be critically important in setting a conceptual framework for developing alternative treatment in ADHD, especially for aerobic exercise intervention. In addition, results of the study contribute to lay the ground work for both scientific and clinical application in adolescents with ADHD.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of ADHD by a board-certified psychiatrist according to the Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-V)
* Adolescents aged between 13-17
* Absence of other neuropsychological disorders including, autism spectrum disorders, mental retardation, psychotic disorders, bipolar disorders, obsessive-compulsive disorder, and neurocognitive disorders
* Right-handed

Exclusion Criteria:

* Presence of other major systematical diseases
* Taking neuropsychological medication within one month, except for medication for ADHD
* With contraindications for non-invasive brain stimulation such as epilepsy, pacemaker or intracranial mental implants
* Color blindness
* Taking part in other studies within one month.

Ages: 13 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 90 (Estimated)
Dates: Start 2023-09-09 (Actual); Primary Completion 2025-10-01 (Estimated); Study Completion 2025-10-01 (Estimated)

PRIMARY OUTCOMES:
Stop Signal Task (SST) | Pre-intervention/immediately after the intervention
  The test will require participants to respond to an arrow stimulus pointing in a given direction. The first set incorporates 16 trials where the participants practice the response. In the second set, the participants will be told to inhibit their response if they heard an auditory signal (a beep). An adaptive staircase will be employed for the stop signal delay allowing the task to adapt to the performance of the participant to result in a 50% success rate. An inter-stimulus interval of 1,000 ms will be applied. The outcome measures are the stop signal reaction time, the estimate of when an individual can successfully inhibit their response 50% of the time. This is inferred as the time before all actions become ballistic, and the person is no longer able to stop the action
Spatial Working Memory (SWM) task | Pre-intervention/immediately after the intervention
  The SWM task is based on a self-ordered search test and assesses primarily nonverbal working memory. Participants are asked to search through a number of colored boxes presented on the screen to find a different token hidden inside. Each box housed only one token per trial. Searching a box more than once during a sequence resulted in within errors, and returning to an emptied box resulted in between errors. A double error could be categorized as both a within and a between error. Two major indices are presented: (1) strategy utilization: the number of search sequences starting with a novel box in both 6- and 8-box problems, and (2) errors in total and three different levels of difficulty (4-, 6-, and 8-box problems): the total errors were calculated as the sum of between errors and within errors minus double errors for searches.
Stockings of Cambridge (SOC) | Pre-intervention/immediately after the intervention
  The SOC requires participants to plan and execute a set of movements to replicate a goal arrangement of balls. At the beginning of each trial, there are two displays shown on the screen simultaneously, and three suspended vertical stockings and three colored balls are presented. Participants are asked to move the colored balls in a single move at a time between the stockings, to correspond to a goal position shown in the top display within a specified number of moves (2, 3, 4, and 5 moves). In the control condition, they are required to follow the ball movements as quickly as possible to provide baseline measures of reaction and movement times, with each trial being an exact replication of their earlier planning moves. Three major indices are presented: (1) number of problems solved in the specified minimum number of moves; (2) mean moves: the number of moves taken in excess of the specified minimum number, but within the maximum allowed
TMS parameters: Motor evoked potential (MEP) | Pre-intervention/immediately after the intervention
  TMS is applied with a figure-of-eight coil with an internal diameter of 70mm connected to a Magstim stimulator (Magstim, Whiteland, Dyfed, UK), which generates a strong, short-lasting magnetic stimulus. It induces an electric current flow in the motor cortex sufficient to activate neurons at the suprathreshold level, shown as MEP of the representational muscle. Surface MEPs is recorded from the right abductor digiti minimi muscle (ADM) with an Ag-AgCl electrode in a belly-tendon montage. The signals will be filtered (2Hz to 2 kHz, sampling rate 5 kHz), amplified, and then stored on a computer via a Power 1401 data acquisition interface (Cambridge Electronic Design, Cambridge, UK).
  The peak-to-peak amplitude of the MEP is defined as the overall response of the ADM induced by stimulating the contralateral motor cortex by TMS. The mean MEP is averaged in at least 15 trials and recorded as milli voltage.
TMS parameters: Resting motor threshold (RMT) | Pre-intervention/immediately after the intervention
  RMT is defined as the minimum TMS intensity that elicits a peak-to-peak MEP of 50~100 microvoltage (μV) in the relaxed muscle in at least three of six consecutive trials. RMT is recorded by the intensity of TMS presented by percentage (0-100%). The higher percentage represents a stronger intensity to elicit RMT.
TMS parameters: Active motor threshold (AMT) | Pre-intervention/immediately after the intervention
  AMT is the minimum intensity eliciting an MEP response of 200~300 microvoltage (μV) during moderate spontaneous background muscle activity (~15% of the maximum muscle strength) in at least three of six consecutive trials. AMT is recorded by the intensity of TMS presented by percentage (0-100%). The higher percentage represents a stronger intensity to elicit AMT.
TMS parameters: Short-interval intracortical inhibition (SICI) and intracortical facilitation (ICF) | Pre-intervention/immediately after the intervention
  In the SICI-ICF protocol, a subthreshold conditioning stimulus (determined as 70 % of AMT) precedes the test stimulus (determined as baseline MEP of ~1mV) with the interstimulus intervals (ISIs) of 2, 3, 5, 10, and 15ms. The first three ISIs reflect inhibitory and the last two ISIs reveal facilitatory effects. The pairs of stimuli are organized into 15 blocks. Each block contains double pulses with all ISIs, and one additional single test pulse in a pseudo-randomized order for each block. SICI is mainly influenced by GABAA receptors and ICF is thought to predominantly reflect the activity of the glutamatergic system, with some GABAA contribution. The SICI-ICF is presented as the subtraction of the conditioning stimulus by the test stimulus.

CONTACTS AND LOCATIONS:
Overall Officials: Hsiao-I Kuo, Ph.D., Principal Investigator — NTUPT
Locations (1):
- Neurophysiology and Cognition in Children and Young Adults Lab, School and Graduate Institute of Physical Therapy of National Taiwan University (NTU-PT), Taipei County, Taiwan

IPD SHARING:
Plan to Share IPD: No